CLINICAL TRIAL: NCT04274426
Title: A Randomized Phase II Trial of Mirvetuximab Soravtansine (IMGN853), in Folate Receptor Alpha (FRα) High Recurrent Ovarian Cancer Eligible for Platinum-based Chemotherapy. Supported by: DIAGNOSTIC PROTOCOL for the VENTANA FOLR1 (FOLR1-2.1) CDx Assay Ventana No. RD004881; Protocol Document No. D152967
Brief Title: Mirvetuximab Soravtansine (IMGN853), in Folate Receptor Alpha (FRα) High Recurrent Ovarian Cancer
Acronym: MIROVA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AGO Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR 2.34; 2018-004207-39 (EudraCT Number)
Record Dates: First submitted 2020-02-10; First posted 2020-02-18 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Epithelial Ovarian, Fallopian or Peritoneal Carcinoma
MeSH Terms: interventions — Carboplatin; liposomal doxorubicin; Gemcitabine; Paclitaxel; mirvetuximab soravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control arm with Platinum-based chemotherapy (Active Comparator): 1. Carboplatin (AUC5, d1) combined with pegylated liposomal doxorubicin (PLD) (30 mg/m², d1) q28d
  2. Carboplatin (AUC4, d1) combined with gemcitabine (1000 mg/m2, d1 & d8) q21d
  3. Carboplatin (AUC5, d1) combined with paclitaxel (175 mg/m², d1) q21d
  Interventions: Drug: Carboplatin; Drug: Pegylated liposomal doxorubicin (PLD); Drug: Gemcitabine; Drug: Paclitaxel
- Carboplatin + Mirvetuximab soravtansine (IMGN853) (Experimental): Carboplatin (AUC5, d1) + Mirvetuximab soravtansine (IMGN853) 6 mg/kg IV d1 x 6 cycles q21d, followed by subsequent monotherapy of Mirvetuximab soravtansine (IMGN853) 6 mg/kg IV q3w until disease progression.
  Interventions: Drug: Carboplatin; Drug: Mirvetuximab Soravtansine

INTERVENTIONS:
Drug: Carboplatin — Carboplatin will administered by intravenous route
Drug: Pegylated liposomal doxorubicin (PLD) — PLD will be administered by intravenous route
  Arms: Control arm with Platinum-based chemotherapy
Drug: Gemcitabine — Gemcitabine will be administered by intravenous route
  Arms: Control arm with Platinum-based chemotherapy
Drug: Paclitaxel — Paclitaxel will be administered by intravenous route
  Arms: Control arm with Platinum-based chemotherapy
Drug: Mirvetuximab Soravtansine — Mirvetuximab Soravtansine will be administered by intravenous route
  Arms: Carboplatin + Mirvetuximab soravtansine (IMGN853)

SUMMARY:
This is a multi-center, randomized, two-arm, open-label, comparative phase II trial of Mirvetuximab soravtansine (IMGN853), in folate receptor alpha (FRα) high recurrent ovarian cancer eligible for platinum-based chemotherapy.

DETAILED DESCRIPTION:
136 patients will be randomized into the follow-ing two treatment arms as specified below:

Arm A: Control arm Platinum-based chemotherapy Arm B: Carboplatin + Mirvetuximab soravtansine (IMGN853)

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have a pathologically documented, definite diagnosis of epithelial cancer of the ovary, the fallopian tube or the peritoneum
2. Relapsed disease with a platinum-free interval >3 months
3. All histologic subtypes of ovarian carcinoma including carcinosarcoma (malignant mixed Mullerian tumors, MMMT)
4. Patients with wildtype BRCA1/2 mutation status or with a deleterious BRCA1/2 mutation in germline or somatic testing if they underwent PARP inhibitor therapy in previous treatment line.
5. Patients must be willing to provide archival tumor tissue from current relapse or previous surgeries/biopsies for central confirmation of FRα high status by PS2+ scoring:

   all tumors must exhibit ≥75% of tumor cells with FRα membrane staining and ≥ 2+ intensity by immunohistochemistry (IHC) using the Ventana FOLR1 (FOLR1 2.1) CDx assay.
6. Patients must have measurable disease or evaluable disease in combination with GCIG CA-125 criteria.
7. Patients had one or more prior lines of chemotherapy. The last line of chemotherapy should have included platinum and has resulted in a partial or complete response.
8. Major surgery (not including placement of vascular access device, tumor punch/scrape biopsies or secondary wound closure) must be completed four weeks prior to Day 1.
9. Patients must have adequate hematological, liver, cardiac and kidney function:

   1. Hemoglobin ≥ 10.0 g/dL.
   2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   3. Platelet count ≥ 100 x 109/L.
   4. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
   5. Aspartate aminotransferase/Serum Glutamic Oxaloacetic Transaminase (ASAT/SGOT)) and Alanine aminotransferase/Serum Glutamic Pyruvate Transaminase (ALAT/SGPT)) ≤ 2.5 x ULN, unless liver metastases are present in which case they must be ≤ 5 x ULN.
   6. Serum creatinine ≤ 1.5 x institutional ULN and glomerular filtration rate of at least 40 ml/minute according to Cockroft-Gault formula.
10. Patient is female and ≥18 years of age at the time of the first screening visit.
11. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
12. Patients must be willing and able to sign the informed consent form, and to adhere to the study visit schedule and other protocol requirements.
13. Women of childbearing potential (a woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently ster-ile. Permanent sterilization methods include hysterectomy, bi-lateral salpingectomy and bilateral oophorectomy) must have a negative serum pregnancy test within 3 days from day 1 of cycle 1 and agree to use a highly effective method of contraception while on study treatment and for at least 6 months after end of treatment. Such methods include:

    1. Combined (estrogen and progestogen containing) hor-monal contraception associated with inhibition of ovulation:

       * oral
       * intravaginal
       * transdermal
    2. Progestogen-only hormonal contraception associated with inhibition of ovulation:

       * oral
       * injectable
       * implantable
    3. Intrauterine device (IUD)
    4. Intrauterine hormone-releasing system ( IUS)
    5. Bilateral tubal occlusion
    6. Vasectomized partner
    7. Sexual abstinence

Exclusion Criteria:

1. Non-epithelial tumor origin of the ovary, the fallopian tube or the peritoneum (i.e. germ cell tumors)
2. Ovarian tumors of low malignant potential (e.g. borderline tumors).
3. Unknown BRCA status.
4. Patients who are planned to receive bevacizumab for the current relapse.
5. Other malignancy within the last 3 years (except cervix or breast in situ carcinoma, type I stage I endometrial cancer)
6. Patients who underwent surgery for the current relapse with macroscopic complete resection
7. Prior systemic anticancer therapy within 28 days before randomization
8. Prior treatment with folate receptor-targeting investigational agents is not allowed.
9. Patients with > Grade 1 peripheral neuropathy.
10. Serious concurrent illness or clinically-relevant active infection
11. Previous clinical diagnosis of non-infectious interstitial lung disease, including non-infectious pneumonitis.
12. Active or chronic corneal disorders such as Sjogren's syndrome, Fuchs corneal dystrophy (requiring treatment), history of corneal transplantation, active herpetic keratitis, active ocular conditions requiring ongoing treatment/monitoring such as uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema, and /or monocular vision. Active or chronic corneal disorder
13. Required use of folate-containing supplements (e.g. folate deficiency)
14. Women of childbearing potential (WOCBP) not protected by highly effective contraceptive methods.
15. Pregnant and/or breast-feeding women.
16. Known hypersensitivity to one of the chemotherapy re-gimes and/or PARP inhibitors and/or any of their excipients.
17. Patients with prior hypersensitivity to monoclonal antibodies.
18. Patients with potential risks according to contraindication, warnings or interactions of the used chemotherapeutic agents as stated in the SmPCs are not eligible for partici-pation in this trial.
19. Patients with untreated or symptomatic central nervous system (CNS) metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) defined as the time from randomization to progressive disease (PD) or death, whichever occurs earlier. PD is based on investigator assess-ment using the Response Evaluation Criteria in Solid Tumors (RECIST 1.1). | Up to 2.5 years. From date of randomization until date of progressive disease (PD) or death, whichever occurs earlier.
  PD is based on investigator assessment using the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

SECONDARY OUTCOMES:
OS | Up to 2.5 years. From date of randomization until date of death from any cause.
  Overall survival
ORR | Up to 2.5 years. From date of randomization to date of death death from any cause.
  Objective response rate
Efficacy regarding PFS | Up to 2.5 years. From date of randomization to date of death from any cause.
  Efficacy regarding Progression Free Survival depending on histologic subtype
Efficacy regarding OS | Up to 2.5 years. From date of randomization to date of death from any cause.
  Efficacy regarding Overall Survival depending on histologic subtype
Efficacy regarding ORR | Up to 2.5 years. From date of randomization to date of death from any cause.
  Efficacy regarding Objective Response Rate depending on histologic subtype
Serological progressive disease | Up to 2.5 years. From date of randomization to date of death death from any cause.
  Time to serological progressive disease according to GCIG criteria
Time to first subsequent treatment (TFST) | Up to 2.5 years. From date of randomization to date of death from any cause.
  Time to first subsequent treatment (TFST)
Time to second subsequent treatment (TSST) | Up to 2.5 years. From date of randomization until date of death from any cause.
  Time to second subsequent treatment (TSST)
Patient-reported outcomes | Up to 2.5 years. From date of randomization until date of death from any cause.
  Quality of Life (EORTC C-30)
Patient-reported outcomes | Up to 2.5 years. From date of randomization until date of death from any cause.
  Quality of Life (EORTC OV28)
Safety and tolerability | Up to 2.5 years. From date of randomization until date of death from any cause through study completion.
  Safety and tolerability of the used drugs evaluated by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Harter, Study Chair — Kliniken Essen-Mitte, Germany
Locations (19):
- Germany (19):
  - Charite Campus Virchow Klinikum, Berlin
  - Städtische Klinikum Dessau, Dessau
  - Universitätsklinikum Carl-Gustav-Carus an der Technischen Universität Dresden, Dresden
  - Evangelische Kliniken-Essen-Mitte, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Mammazentrum HH am Krankenhaus Jerusalem, Hamburg
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - ViDia Christliche Kliniken Karlsruhe, Karlsruhe
  - St. Elisabeth-Krankenhaus GmbH, Köln-Hohenlind
  - HELIOS Klinikum Krefeld, Krefeld
  - Klinikum Mannheim, Mannheim
  - OnkoNet Marburg, Marburg
  - Klinikum der Universität München, München
  - Rotkreuzklinikum München, München
  - TU München, Klinikum recht der Isar, München
  - Universitätsklinik Münster, Münster
  - Klinikum Südstadt Rostock, Rostock
  - Universitätsfrauenklinik Ulm, Ulm

REFERENCES:
- See also: Related Info — http://www.ago-ovar.de/